CLINICAL TRIAL: NCT06674096
Title: Rituximab，Lenalidomide and Chidamide Followed by CR-CHOP in Elderly Patients with Newly-diagnosed Double-expressor Lymphoma
Brief Title: RLC Followed by CR-CHOP in Elderly Patients with Newly-diagnosed DEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Chief director of Lymphoma Department, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLC-CRCHOP
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Double-expressor Lymphoma
Keywords: DLBCL; DEL; rituximab; lenalidomide; chidamide; chemo-free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RLC-CRCHOP (Experimental): Introduction treatment: Rituximab, lenalidomide, chidamide for 2 cycles:
  rituximab 375mg/m2, d1, lenalidomide 10mg qd d1-14, chidamide 20mg, d1,4,8,11.
  Immunochemtherapy phase: CR CHOP for 4 cycles: chidamide 20mg d1,4,8,11,rituximab 375mg/m2 d0, cyclophosphamide: 750mg/m2 d1, epirubicin: 75mg/ m2 d1 (or liposomal doxorubicin 35mg/m2 d1), vindesine 4mg d1, prednisone: 100mg, d1-5.
  maintenance treatment period: chidamide d1,4,8,11
  Interventions: Drug: RLC-CRCHOP

INTERVENTIONS:
Drug: RLC-CRCHOP — Introduction treatment: Rituximab, lenalidomide, chidamide for 2 cycles:
  rituximab 375mg/m2, d1, lenalidomide 10mg qd d1-14, chidamide 20mg, d1,4,8,11.
  Immunochemtherapy phase: CR CHOP for 4 cycles: chidamide 20mg d1,4,8,11,rituximab 375mg/m2 d0, cyclophosphamide: 750mg/m2 d1, epirubicin: 75mg/ m2 d1 (or liposomal doxorubicin 35mg/m2 d1), vindesine 4mg d1, prednisone: 100mg, d1-5.
  maintenance treatment period: chidamide d1,4,8,11

SUMMARY:
This is a prospective, single-arm, multicenter clinical study to evaluate the efficacy and safety of chidamide, rituximab combined with lenalidomide sequential immunochemotherapy in the treatment of newly diagnosed elderly double-expressor diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
It is divided into 4 stages: screening period, induction therapy period, immunochemotherapy period and maintenance therapy period. The screening period was 28 days before the first dose. Introduction treatment period: Enrolled subjects received RLC regimen every 21 days for a cycle of 2 cycles. Immunochemotherapy phase: CR-miniCHOP regimen was administered after the completion of the introduction therapy phase. Every 21 days for a cycle, treatment for 4 cycles. Patients who achieved CR with induction therapy entered the maintenance treatment period, receiving 20 mg of chidamide d1,4,8,11 recommended 8 cycles. Patients who did not achieve CR were discontinued from the study and treated at the discretion of their physician.

ELIGIBILITY:
Inclusion Criteria:

* 1. Untreated DLBCL patients confirmed by histopathology 2. Immunohistochemistry showed positive expression of MYC and BCL2 protein (double expressor lymphoma, MYC≥40%, BCL2≥50%) 3. age over 70 years old or age ≥65 years old and ECOG score ≥2 points, both male and female 4. Having at least one evaluable lesion, defined as having at least one lymphadenopathy with a maximum diameter > 1.5 cm, or at least one extranodal lesion with a maximum diameter > 1.0 cm, and at least two vertical diameters that can be accurately measured.

  5. ECOG PS≤3 6. Expected survival time ≥3 months 7. voluntary participation in clinical research; Fully understand and understand the study and sign the informed consent; Willingness to follow and ability to complete all research steps.

Exclusion Criteria:

* 1. The pathological subtypes were PCNSL, PMBCL, EBV-positive DLBCL and HGBL 2. Hemophagocytic syndrome accompanied the diagnosis 3. Central nervous system involvement is secondary to lymphoma 4. Are participating in other clinical studies, or the first study drug is administered less than 4 weeks after the end of treatment in the previous clinical study 5. HIV infection 6. Major surgery was performed within 28 days prior to study start 7. Any active infection that required systematic anti-infective therapy developed within 14 days prior to study initiation 8. The patients considered by the investigator to be unsuitable for participating in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-06 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of first day of treatment until the date of first documented date of disease progression or death from any cause, assessed up to 24 months
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | 21days after the end of treatment
  overall response rate
CRR | 21days after the end of treatment
  complete response rate
OS | : From date of first day of treatment until the date of first documented date of death from any cause, assessed up to 24 months
  Overall Survival
AE and SAE | From date of first day of treatment until 30 day after last treatment
  Adverse event and serious adverse event
Performance status | At screening period, after 2 cycles of ZR2 regimen(each cycle is 21 days), after 2 cycles of RCHOP regimen(each cycle is 21 days) and 21days after the end of treatment
  Assess the patient's performance status according to the Barthel index. Patients will be classified into 5 scales with the score ranging from 0 to 100: 0-20 points=extremely severe functional impairment; 25-45 points=severe functional impairment; 50-70 points=moderate functional impairment; 75-95 points=mild functional impairment; 100 points=normal. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No